CLINICAL TRIAL: NCT01499004
Title: A Phase 1, Randomized, Open Label, Partial Crossover Study To Evaluate The Pharmacokinetics (PK) And Safety Of Three Modified Release (MR) And One Immediate Release (IR) Formulations Of Tofacitinib (CP-690,550) In Healthy Volunteers
Brief Title: A Phase 1 Study To Evaluate The Pharmacokinetics And Safety Of Three Modified Release And One Immediate Release Formulations Of Tofacitinib (CP-690,550) In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A3921131
Record Dates: First submitted 2011-11-23; First posted 2011-12-26 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: tofacitinib; CP-690; 550; relative bioavailability; modified release; Phase 1
MeSH Terms: interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment A (Experimental): tofacitinib (CP-690,550) modified-release formulation A-Fed
  Interventions: Drug: tofacitinib (CP-690,550) modified-release formulation A
- Treatment B (Experimental): tofacitinib (CP-690,550) modified-release formulation B1-Fed
  Interventions: Drug: tofacitinib (CP-690,550) modified-release formulation B1
- Treatment C (Experimental): tofacitinib (CP-690,550) modified-release formulation A-Fasted
  Interventions: Drug: tofacitinib (CP-690,550) modified-release formulation A
- Treatment D (Experimental): tofacitinib (CP-690,550) modified-release formulation B1-Fasted
  Interventions: Drug: tofacitinib (CP-690,550) modified-release formulation B1
- Treatment E (Experimental): tofacitinib (CP-690,550) modified-release formulation B2-Fasted
  Interventions: Drug: tofacitinib (CP-690,550) modified-release formulation B2
- Treatment F (Experimental): tofacitinib (CP-690,550) immediate-release formulation-Fasted
  Interventions: Drug: tofacitinib (CP-690,550) immediate-release formulation

INTERVENTIONS:
Drug: tofacitinib (CP-690,550) modified-release formulation A — A single dose of 22 mg tofacitinib (CP-690,550) modified-release formulation A administered with food.
  Arms: Treatment A
Drug: tofacitinib (CP-690,550) modified-release formulation B1 — A single dose of 22 mg tofacitinib (CP-690,550) MR-B1 formulation administered with food
  Arms: Treatment B
Drug: tofacitinib (CP-690,550) modified-release formulation A — A single dose of 22 mg tofacitinib (CP-690,550) modified-release formulation A administered without food
  Arms: Treatment C
Drug: tofacitinib (CP-690,550) modified-release formulation B1 — A single dose of 22 mg tofacitinib (CP-690,550) modified-release formulation B1 administered without food
  Arms: Treatment D
Drug: tofacitinib (CP-690,550) modified-release formulation B2 — A single dose of 22 mg tofacitinib (CP-690,550) modified-release formulation B2 administered without food
  Arms: Treatment E
Drug: tofacitinib (CP-690,550) immediate-release formulation — A single dose of 10 mg tofacitinib (CP-690,550) immediate-release formulation administered without food
  Arms: Treatment F

SUMMARY:
This study will explore the drug behavior and safety following a single dose of three different 22 milligram tofacitinib (CP-690,550) modified-release formulations in 30 healthy volunteers. These formulations will be compared to 10 milligram tofacitinib (CP-690-550) in an immediate-release formulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects and/or healthy females subjects who are of non-childbearing potential.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease;
* Clinically significant infections within the past 3 months

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
AUCinf: Area under the plasma concentration-time profile from time 0 exprapolated to infinite time | 72 hours post dose
AUClast: Area under the plasma concentration-time profile from time 0 to the last with quantifiable concentration | 72 hours post dose
Cmax: Maximum plasma concentration of tofacitinib (CP-690,550) | 72 hours post dose
Tmax: Amount of time tofacitinib (CP-690,550) is at maximum plasma concentration | 72 hours post dose
t1/2: The time required for one half of the total amount of tofacitinib (CP-690,550) to be removed from the plasma | 72 hours post dose

SECONDARY OUTCOMES:
Frel: Relative bioavailability (Frel) of tofacitinib (CP-690,550) in the modified-release formulations compared to the immediate release formulation | 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921131&StudyName=A%20Phase%201%20Study%20To%20Evaluate%20The%20Pharmacokinetics%20And%20Safety%20Of%20Three%20Modified%20Release%20And%20One%20Immediate%20Release%20Formulations%20Of%20Tofaci